CLINICAL TRIAL: NCT03177005
Title: Expanded Access for Hereditary Angioedema (HAE)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Joshua S. Jacobs, MD (Industry)
Responsible Party: Sponsor-Investigator, Joshua S. Jacobs, MD, Treating HCP, CSL Behring
Organization: CSL Behring (Industry)
Other Study IDs: CSL830
Record Dates: First submitted 2017-05-30; First posted 2017-06-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: CSL830

SUMMARY:
Approval for access is solely at CSL Behring's discretion and the following criteria must be met for CSL Behring to consider access to experimental or unlicensed product:

* The patient has an unmet medical need that is life-threatening, chronic or seriously disabling, as defined by local regulations and applicable to the particular patient. All treatment options available to the patient should have been explored and exhausted by the physician, including participation in clinical trials.
* The patient and caregiver must be informed of potential risks and benefits of receiving the experimental therapy. The overall potential benefit should outweigh the combined potential risks of the experimental medicine and the outcome of the illness or disease itself. If approved, CSL Behring will provide treating physicians with risk information wording for inclusion in the physician's informed consent form, which will outline the risks of the experimental medicine. Treating physicians must share this information with the patient through the informed consent process. Treating physicians must also agree to participate in CSL Behring's safety monitoring and reporting requirements and follow FDA safety reporting regulations.
* Only medicines under active clinical development in the USA by CSL Behring will be considered for early access. There must be sufficient clinical trial data on efficacy and safety indicating a potential benefit greater than risks for the intended use and dose.
* Granting early access should not negatively impact or delay the ongoing development program with the experimental medicine to support approval by FDA and other regulatory authorities.
* Adequate supply of the experimental medicine must exist to support both ongoing clinical trials and approved expanded access until, and if, the product becomes commercially available.

Only requests received from the licensed physician on behalf of the patient will be considered. CSL Behring will assess the request against the above criteria. If these criteria are met and the IRB/Ethics Committee and FDA approve access to the experimental therapy, early access may be granted. US medicine importation requirements must also be met. The patient's physician is responsible for the patient's ongoing care as well as all relevant US federal and state legislations while the patient is receiving the experimental medicine through early access. If approved the patient/caregiver must provide informed consent and the treating physician must follow safety and monitoring requirements as defined by CSL Behring.

CSL Behring cannot provide a guarantee that expanded access will be available for every experimental medicine. Even if such a program is offered CSL Behring cannot guarantee that an experimental medicine will be available to a particular patient. The early access will cease if clinical trials or regulatory assessment determines the product does not demonstrate a positive risk benefit for patients. Once the experimental medicine is approved and commercially available in the US, early access will no longer be available.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

REFERENCES:
- See also: CSL Behring's Expanded Access Program — http://www.cslbehring-us.com/healthcare-professionals/expanded-access-program.htm